CLINICAL TRIAL: NCT00403832
Title: Comparison of Two Different Acrylate Intraocular Lenses in Cataract Surgery in Patients With Non-infectious Uveitis
Brief Title: Acrylate Intraocular Lenses in Cataract Surgery of Uveitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Franziskus Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-2911
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2009-08

CONDITIONS: Uveitis; Cataract
MeSH Terms: conditions — Uveitis; Cataract

INTERVENTIONS:
Device: intraocular lenses: Two foldable, acrylic, sharp edged IOLs: AcrySof™ (AcrySof SA60AT, Alcon), and Akreos adapt™ (Bausch & Lomb)

SUMMARY:
Cataract is a common complication in uveitis patients. Cataract operations with intraocular lens implantation are difficult in these patients because of complication due to the biocompatibility of the intraocular lens. In this study, uveal and capsular biocompatibility of two widely used acrylate intraocular lenses are compared.

ELIGIBILITY:
Inclusion Criteria:

* non infectious uveitis
* no active inflammation
* significant visual disturbance related to lens opacification

Exclusion Criteria:

* vitreous opacification
* ocular hypertension/glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-08; Study Completion 2007-02

PRIMARY OUTCOMES:
visual acuity
cell deposits on anterior IOL surface
posterior capsular opacification

CONTACTS AND LOCATIONS:
Overall Officials: Arnd Heiligenhaus, Md Phd, Principal Investigator — Department of Ophthalmology at St.-FranziskusHospital Münster
Locations (1):
- Department of Ophthalmology at St.-Franziskus Hospital, Münster, Germany

REFERENCES:
- [Derived] Roesel M, Heinz C, Koch JM, Heiligenhaus A. Comparison of orbital floor triamcinolone acetonide and oral prednisolone for cataract surgery management in patients with non-infectious uveitis. Graefes Arch Clin Exp Ophthalmol. 2010 May;248(5):715-20. doi: 10.1007/s00417-009-1269-1. Epub 2010 Jan 16. PMID 20082200
- See also: Related Info — http://www.uveitis-zentrum.de